CLINICAL TRIAL: NCT00547950
Title: A Model Study on the Comprehensive Treating Protocol of Secondary Prevention and Effect Evaluation of Ischemic Stroke With Traditional Chinese Medicine
Brief Title: A Multiple-Centered, Prospective Cohort Study: the Second Prevention Trial for Ischemic Stroke With Deng Zhan Sheng Mai Capsule（SPIRIT-DZSM-2）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006BAI04A02-2
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): drug
  Interventions: Drug: :Deng Zhan Sheng Mai Capsule

INTERVENTIONS:
Drug: :Deng Zhan Sheng Mai Capsule — capsule，0.18g，2＃，po，Bid*1year.

SUMMARY:
In order to observe the influence of the Dengzhan Shengmai Capsule on the endpoint of patients with ischemic stroke, we hold the multi-centered prospective cohort study. From November 2007 to December 2009, 12000 subjects are included in 200 clinical research centers all over China. The subjects naturally formed two cohorts based on taking Dengzhan Shengmai capsule or not. The basic therapy included antiplatelet aggregation , stroke health education, management of blood pressure, blood lipid and blood glucose, etc. Then all of the subjects are visited on the 360th day after inclusion. The recurrence of stroke, cardiovascular events, and peripheral arterial events are observed.

ELIGIBILITY:
Inclusion Criteria:

* 40-75 years old
* Ischemic stroke diagnosed by CT/MRI scan
* Patient presenting from 14 days to 6 months of first onset of Ischemic stroke.
* Presence of at least one risk factor of stroke (such as hypertension, Diabetes mellitus, coronary heart disease, hyperlipidemia, and smoking, etc.)that can be interfered in.
* Informed consent.

Exclusion Criteria:

* Silent cerebral infarction;
* Patients after vasculoplasty with Intracranial Artery Stenosis.
* Watian drinking test≥grade 4.
* MRS=grade 5.
* Cerebral infarction due to other causes except arterial Sclerosis(i.e. cardiogenic embolism, arteritis, polycythemia vera, primary thrombocythemia, sickle-cell anemia,, thrombotic thrombocytopenia purpura, DIC, cerebral amyloid angiopathy, Moyamoya disease, intracranial vascular malformations etc);
* Presence of serious heart disease, heart, liver, lung, and kidney functional failure; malignancy; alimentary tract hemorrhage;
* Patients with mental disorder.
* Patients that cannot take medicine due to other causes
* Females during pregnancy or lactation.
* Already attend other clinical trial.
* That unsuitable for clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2007-11; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
recurrence of stroke | 1 year

SECONDARY OUTCOMES:
Cardiovascular events and other peripheral vascular events Modified Rankin Scale (mRS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yan Huang, Bachelor, Principal Investigator — Guangdong Province Hospital of Tradtional Chinese Medicine
Locations (1):
- Guangdong Province Hospital of Tradtional Chinese Medicine, Guangzhou, Guangdong, China